CLINICAL TRIAL: NCT01871545
Title: Evaluation of HCC Response to Systemic Therapy With Quantitative MRI
Brief Title: Evaluation of Liver Cancer With Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Bachir Taouli, Professor, Radiology and Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 12-0214
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Hepatocellular Carcinoma; HCC
Keywords: hepatocellular carcinoma; HCC; liver cancer; liver disease; magnetic resonance imaging; MRI
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Liver Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnetic Resonance Imaging (Experimental): dynamic contrast-enhanced MRI measuring arterial and portal flow
  Interventions: Device: Magnetic Resonance Imaging
- Healthy Controls (No Intervention)

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Magnetic Resonance Imaging is a radiation free non invasive technique using magnetic radiofrequency waves to image the body. In this study, the research team would like to investigate the possibility of providing functional information on aggressiveness, vascularity and oxygen uptake in liver cancer tumors.
  Other Names: MRI
  Arms: Magnetic Resonance Imaging

SUMMARY:
The incidence of hepatocellular carcinoma (HCC) has recently increased in the United States. Although imaging plays a major role in HCC screening and staging, the possibility of predicting HCC tumor grade, aggressiveness, angiogenesis and hypoxia with imaging are unmet needs. In addition, new antiangiogenic drugs now available to treat advanced HCC necessitate the use of new imaging criteria beyond size. The investigators would like to develop and validate non-invasive magnetic resonance imaging (MRI) methods based on advanced diffusion-weighted imaging (DWI), MR Elastography, BOLD (blood oxygen level dependent) MRI and perfusion-weighted imaging (PWI, using gadolinium contrast) to be used as non-invasive markers of major histopathologic features of HCC, and to predict and assess early response of HCC to systemic therapy. The investigators also would like to develop quality control tools to improve the quality and decrease variability of quantitative MRI metrics. These techniques combined could represent non-invasive correlates of histologic findings in HCC, could enable individualized therapy, and provide prognosis in patients with HCC.

DETAILED DESCRIPTION:
The incidence of hepatocellular carcinoma (HCC) has recently increased in the US mostly due to an increase in chronic hepatitis C infection. Angiogenesis is critical for the growth and metastatic progression of HCC. With the development of new antiangiogenic drugs such as sorafenib, imaging methods to predict and assess therapeutic response beyond changes in size become critical. However, validated imaging methods to predict and assess early HCC response to targeted agents are lacking.

In this study, the investigators would like to develop quantitative MRI methods interrogating different features of HCC tumor biology and pathology, including tumor cellularity, grade, angiogenesis and hypoxia. The investigators propose a multiparametric approach combining advanced DWI (IVIM: intravoxel incoherent motion diffusion measuring perfusion fraction and true diffusion coefficient), DCE-MRI (dynamic contrast-enhanced MRI, which measures arterial and portal flow, mean transit time, blood volume and distribution volume), and BOLD MRI using oxygen or carbogen challenge. This protocol will be performed in patients with HCC undergoing hepatic resection. Routine and advanced histopathologic methods will be performed (tumor grade, CK19 expression, presence of microvascular invasion, VEGF expression, microvessel density, HIF 1-alpha expression). MRI metrics will be correlated with histopathologic metrics.

The first portion of the proposal involves the development of a QC algorithm assessing MR data quality and test-retest. The investigators will propose solutions to improve data acquisition and processing. The last 2 years of the study will be dedicated to a prospective randomized study comparing Yttrium 90 radioembolization to sorafenib, assessing the role of baseline MRI metrics and early changes (at 2 weeks) in these metrics as markers of tumor response and time to progression in patients with unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

Study group

* Patients diagnosed with HCC, who will undergo resection or transplantation within 6 months, as part of routine clinical care and patients diagnosed with unresectable HCC
* 18 years of age and older
* Patient is able to give informed consent for this study

Control group

* Healthy volunteers 18 years of age and older
* Subject is able to give informed consent for this study

Exclusion Criteria:

* Age less than 18 years
* Unable or unwilling to give informed consent
* Contra-indications to MRI:

  1. Electrical implants such as cardiac pacemakers or perfusion pumps
  2. Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
  3. Ferromagnetic objects such as jewelry or metal clips in clothing
  4. Pregnant subjects
  5. Pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-06; Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bachir Taouli, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment from June 2013 through February 2018
Groups:
- Hepatocellular Carcinoma (HCC): Participant with hepatocellular carcinoma (HCC)
- Healthy Volunteer: Healthy volunteer participant
Period: Overall Study
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Volunteer
Started | 73 | 11
Completed | 56 | 8
Not Completed | 17 | 3
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 11 | 2
Not completed — Physician Decision | 4 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Hepatocellular Carcinoma (HCC): Participants with hepatocellular carcinoma (HCC)
- Healthy Participant: Healthy control participants
- Total: Total of all reporting groups
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant | Total
Number analyzed (Participants) | 56 | 8 | 64
Age, Continuous [Median (Full Range); unit: years] | 65 [23 to 93] | 36 [23 to 55] | 62 [23 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 44 | 1 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 1 | 18
  Not Hispanic or Latino | 36 | 7 | 43
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 1 | 19
  White | 31 | 4 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
SubStudy 1: Age [Median (Full Range); unit: years] — Population: Data analysis only for a subset of patients with HCC undergoing hepatic resection compared to healthy controls.
  years
    number analyzed (Participants) | 32 | 8 | 40
    (all) | 59 [30 to 71] | 36 [23 to 55] | 59 [30 to 71]
SubStudy 1: Sex [Count of Participants; unit: Participants] — Population: Data analysis only for a subset of patients with HCC undergoing hepatic resection compared to healthy controls.
  Participants
    number analyzed (Participants) | 32 | 8 | 40
    Female | 6 | 7 | 13
    Male | 26 | 1 | 27
SubStudy 1: Ethnicity [Count of Participants; unit: Participants] — Population: Data analysis only for a subset of patients with HCC undergoing hepatic resection compared to healthy controls.
  Participants
    Hispanic or Latino: number analyzed (Participants) | 32 | 8 | 40
    Hispanic or Latino | 7 | 1 | 8
    Not Hispanic or Latino: number analyzed (Participants) | 32 | 8 | 40
    Not Hispanic or Latino | 24 | 7 | 31
    Unknown or Not Reported: number analyzed (Participants) | 32 | 8 | 40
    Unknown or Not Reported | 1 | 0 | 1
SubStudy 1: Race [Count of Participants; unit: Participants] — Population: Data analysis only for a subset of patients with HCC undergoing hepatic resection compared to healthy controls.
  Participants
    American Indian or Alaska Native: number analyzed (Participants) | 32 | 8 | 40
    American Indian or Alaska Native | 0 | 0 | 0
    Asian: number analyzed (Participants) | 32 | 8 | 40
    Asian | 3 | 3 | 6
    Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 32 | 8 | 40
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American: number analyzed (Participants) | 32 | 8 | 40
    Black or African American | 12 | 1 | 13
    White: number analyzed (Participants) | 32 | 8 | 40
    White | 16 | 4 | 20
    More than one race: number analyzed (Participants) | 32 | 8 | 40
    More than one race | 0 | 0 | 0
    Unknown or Not Reported: number analyzed (Participants) | 32 | 8 | 40
    Unknown or Not Reported | 1 | 0 | 1
SubStudy 2: Age [Median (Full Range); unit: years] — Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
  years
    number analyzed (Participants) | 24 | 0 | 24
    (all) | 68 [55 to 93] |  | 68 [55 to 93]
SubStudy 2: Sex [Count of Participants; unit: Participants] — Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
  Participants
    number analyzed (Participants) | 24 | 0 | 24
    Female | 6 |  | 6
    Male | 18 |  | 18
SubStudy 2: Ethnicity [Count of Participants; unit: Participants] — Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
  Participants
    Hispanic or Latino: number analyzed (Participants) | 24 | 0 | 24
    Hispanic or Latino | 10 |  | 10
    Not Hispanic or Latino: number analyzed (Participants) | 24 | 0 | 24
    Not Hispanic or Latino | 12 |  | 12
    Unknown or Not Reported: number analyzed (Participants) | 24 | 0 | 24
    Unknown or Not Reported | 2 |  | 2
SubStudy 2: Race [Count of Participants; unit: Participants] — Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
  Participants
    American Indian or Alaska Native: number analyzed (Participants) | 24 | 0 | 24
    American Indian or Alaska Native | 0 |  | 0
    Asian: number analyzed (Participants) | 24 | 0 | 24
    Asian | 1 |  | 1
    Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 24 | 0 | 24
    Native Hawaiian or Other Pacific Islander | 0 |  | 0
    Black or African American: number analyzed (Participants) | 24 | 0 | 24
    Black or African American | 6 |  | 6
    White: number analyzed (Participants) | 24 | 0 | 24
    White | 15 |  | 15
    More than one race: number analyzed (Participants) | 24 | 0 | 24
    More than one race | 0 |  | 0
    Unknown or Not Reported: number analyzed (Participants) | 24 | 0 | 24
    Unknown or Not Reported | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: SubStudy 1: Apparent Diffusion Coefficient (ADC)
Description: Tumor diffusion (apparent diffusion coefficient) measured with diffusion-weighted imaging sequence
Time Frame: Day 1
Population: Data analysis only for a subset of patients with HCC undergoing hepatic resection
Measure: Mean (Standard Deviation); unit: 1x10^-3 mm^2/s
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 32 | 0
1x10^-3 mm^2/s | 1.43 (0.68) |

2. Primary Outcome: SubStudy 1: Total Tumor Perfusion (Ft)
Description: Perfusion/flow measured with dynamic contrast-enhanced imaging using gadolinium contrast
Time Frame: Day 1
Population: Data analysis only for a subset of patients with HCC undergoing hepatic resection
Measure: Mean (Standard Deviation); unit: ml/min/100g
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 32 | 0
ml/min/100g | 358 (337) |

3. Primary Outcome: SubStudy 1: Tumor Arterial Perfusion Fraction (ART)
Description: Perfusion/flow measured with dynamic contrast-enhanced imaging using gadolinium contrast
Time Frame: Day 1
Population: Data analysis only for a subset of patients with HCC undergoing hepatic resection
Measure: Mean (Standard Deviation); unit: percent of perfusion
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 32 | 0
percent of perfusion | 78.9 (21.5) |

4. Primary Outcome: SubStudy 1: Tumor Mean Transit Time (MTT)
Description: Tumor mean transit time (MTT) of contrast agent. Perfusion/flow measured with dynamic contrast-enhanced imaging using gadolinium contrast
Time Frame: Day 1
Population: Data analysis only for a subset of patients with HCC undergoing hepatic resection
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 32 | 0
sec | 21.2 (15.8) |

5. Primary Outcome: SubStudy 1: Tumor Distribution Volume (DV)
Description: Tumor distribution volume (DV) of contrast agent. Perfusion/flow measured with dynamic contrast-enhanced imaging using gadolinium contrast
Time Frame: Day 1
Population: Data analysis only for a subset of patients with HCC undergoing hepatic resection
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 32 | 0
percent | 34.6 (24.7) |

6. Primary Outcome: SubStudy 1: Oxygen Uptake
Description: Oxygen uptake measured with T2* and T1-weighted imaging
Time Frame: Day 1
Population: Data analysis only for a subset of patients with HCC undergoing hepatic resection compared to healthy controls. Oxygen uptake for HCCs is reported in patients, and oxygen uptake for the liver is reported in volunteers. R1 measurements method in the volunteers proved unreliable - therefore no data available for T1/R1 in the healthy participant arm.
Measure: Mean (Standard Deviation); unit: s-1
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 32 | 8
s-1
  R2*(=1/T2*) pre oxygen (O2) administration | 34.6 (24.7) | 33.2 (5.8)
  R2* post O2 | 33.7 (14.5) | 30.7 (5.2)
  ΔR2*=R2* post O2-R2* pre O2: number analyzed (Participants) | 32 | 0
  ΔR2*=R2* post O2-R2* pre O2 | -0.78 (8.7) |
  R1(=1/T1) pre oxygen (O2) administration: number analyzed (Participants) | 32 | 0
  R1(=1/T1) pre oxygen (O2) administration | 1.67 (0.94) |
  R1 post O2: number analyzed (Participants) | 32 | 0
  R1 post O2 | 1.90 (1.79) |
  ΔR1=R1 post O2-R1 pre O2: number analyzed (Participants) | 32 | 0
  ΔR1=R1 post O2-R1 pre O2 | 0.23 (1.1) |

7. Primary Outcome: SubStudy 1: Percent Change in Oxygen Uptake
Description: Oxygen uptake measured with T2* and T1-weighted imaging. Oxygen uptake (% change pre and post O2 administration) calculated by Liver ΔR2*=100 x (R2* post O2-R2* pre O2)/R2* pre O2. The healthy participants breathed 100% medical O2 through a mask for 10 min., and were imaged before and after O2 administration with the MRI methods that are sensitive to oxygen uptake in tumors.
Time Frame: Day 1, pre-oxygen administration and 10 min. post-oxygen administration
Population: Healthy Participants only
Measure: Mean (Standard Deviation); unit: percent of oxygen uptake
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 0 | 8
percent of oxygen uptake |  | 7.2 (7.9)

8. Primary Outcome: SubStudy 2: ADC
Description: Tumor diffusion measured with diffusion-weighted imaging sequence. In diffusion weighted MR imaging (DWI), the signal is proportional to the Brownian motion diffusion of free water protons in tissues. Deposition of collagen in tissue (as in fibrotic disease), or cellularity in tumors act as impediments to free water diffusion. Using different mathematical models, the degree of diffusion can be quantified from the MRI signal, to provide information on diffusion restriction due to disease. From mono exponential fit of diffusion signal, one can obtain the apparent diffusion coefficient (ADC). However, this coefficient reflects free water proton diffusion, as well as transport of water protons in the capillary vessels (capillary perfusion).
Time Frame: baseline and 6 weeks after Y90
Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
Measure: Mean (Standard Deviation); unit: 1x10^-3 mm^2/s
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 24 | 0
1x10^-3 mm^2/s
  Baseline | 1.28 (0.22) |
  6 weeks post y90 | 1.62 (0.24) |

9. Primary Outcome: SubStudy 2: Diffusion Coefficient D
Description: Tumor diffusion measured with diffusion-weighted imaging sequence. To separate the diffusion effect from capillary perfusion, a bi-exponential model is used, which provides 3 coefficients: one is the true diffusion coefficient D, reflecting free water proton diffusion.
Time Frame: baseline and 6 weeks after Y90
Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
Measure: Mean (Standard Deviation); unit: 1x10^-3 mm^2/s
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 24 | 0
1x10^-3 mm^2/s
  Baseline | 1.12 (0.19) |
  6 weeks post y90 | 1.33 (0.23) |

10. Primary Outcome: SubStudy 2: Pseudodiffusion Coefficient D*
Description: Tumor diffusion measured with diffusion-weighted imaging sequence. To separate the diffusion effect from capillary perfusion, a bi-exponential model is used, which provides 3 coefficients: one is the pseudo-diffusion coefficient D*, affected by free diffusion and capillary perfusion.
Time Frame: baseline and 6 weeks after Y90
Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
Measure: Mean (Standard Deviation); unit: 1x10^-3 mm^2/s
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 24 | 0
1x10^-3 mm^2/s
  Baseline | 41.16 (35.73) |
  6 weeks post y90 | 30.1 (14.99) |

11. Primary Outcome: SubStudy 2: Perfusion Fraction (PF)
Description: Tumor diffusion measured with diffusion-weighted imaging sequence. To separate the diffusion effect from capillary perfusion, a bi-exponential model is used, which provides 3 coefficients: one is the perfusion fraction PF, which reflects how much the diffusion-weighted signal is affected by capillary perfusion. PF is a measure of vascularity in the tissue.
Time Frame: baseline and 6 weeks after Y90
Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
Measure: Mean (Standard Deviation); unit: 1x10^-3 mm^2/s
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 24 | 0
1x10^-3 mm^2/s
  Baseline | 22.9 (11.57) |
  6 weeks post y90 | 21.9 (9.43) |

12. Secondary Outcome: SubStudy 2: Total Tumor Perfusion (Ft)
Description: Perfusion/flow measured with dynamic contrast-enhanced imaging using gadolinium contrast
Time Frame: baseline and 6 weeks after Y90
Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
Measure: Mean (Standard Deviation); unit: ml/min/100g tissue
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 24 | 0
ml/min/100g tissue
  Baseline | 64.44 (52.77) |
  6 weeks post y90: number analyzed (Participants) | 21 | 0
  6 weeks post y90 | 49.12 (58.59) |

13. Secondary Outcome: SubStudy 2: Tumor Arterial Perfusion Fraction (ART)
Description: Perfusion/flow measured with dynamic contrast-enhanced imaging using gadolinium contrast
Time Frame: baseline and 6 weeks after Y90
Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
Measure: Mean (Standard Deviation); unit: percent of perfusion
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 24 | 0
percent of perfusion
  Baseline | 76.92 (16.87) |
  6 weeks post y90: number analyzed (Participants) | 21 | 0
  6 weeks post y90 | 52.17 (24.53) |

14. Secondary Outcome: SubStudy 2: Tumor Mean Transit Time (MTT) of Contrast Agent
Description: Perfusion/flow measured with dynamic contrast-enhanced imaging using gadolinium contrast
Time Frame: baseline and 6 weeks after Y90
Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 24 | 0
sec
  Baseline | 27 (13.01) |
  6 weeks post y90: number analyzed (Participants) | 21 | 0
  6 weeks post y90 | 27.86 (12.05) |

15. Secondary Outcome: SubStudy 2: Extravascular Extracellular Volume ve
Description: Perfusion/flow measured with dynamic contrast-enhanced imaging using gadolinium contrast. Extravascular extracellular volume fraction ve (%) - represents the portion of tissue occupied by the extravascular extracellular volume (interstitial space), in which MRI contrast agent can distribute.
Time Frame: baseline and 6 weeks after Y90
Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
Measure: Mean (Standard Deviation); unit: percent of perfusion
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 24 | 0
percent of perfusion
  Baseline | 16.77 (6.44) |
  6 weeks post y90: number analyzed (Participants) | 21 | 0
  6 weeks post y90 | 10.27 (7.39) |

16. Secondary Outcome: Substudy 2: Tumor Stiffness
Description: measured with magnetic resonance elastography
Time Frame: baseline and 6 weeks after Y90
Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization. Excluded: 3 treated with other therapies, 2 deceased before 6 weeks follow-up.
Measure: Mean (Standard Deviation); unit: kilo Pascals (kPa)
Arm/Group | Hepatocellular Carcinoma (HCC) | Healthy Participant
Number analyzed (Participants) | 24 | 0
kilo Pascals (kPa)
  Baseline | 5.0 (2.5) |
  6 weeks post y90: number analyzed (Participants) | 19 | 0
  6 weeks post y90 | 7.0 (3.8) |

17. Secondary Outcome: Tumor Response
Description: Tumor response to treatment is evaluated clinically by radiologists according to RECIST and modified RECIST criteria, by which the diameter of the tumor portion that enhances (lights up on imaging) after administration of gadolinium contrast agent is measured before and after treatment. The response is not reported as diameter or diameter difference in mm, but rather as a qualitative variable: complete response, partial response, stable disease and progressive disease. Complete response means no enhancing tumor regions after treatment (i.e. complete tumor necrosis, no more vascular regions of the tumor that take up contrast), partial response is a decrease in the diameter of the enhancing region, stable disease is unchanged diameter, and progressive disease is an increase in the diameter of the enhancing region after treatment.
Time Frame: 6 weeks and 6-12 months
Population: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Groups:
- Hepatocellular Carcinoma (HCC) at 6 Weeks: Participants with hepatocellular carcinoma (HCC) looking at 25 lesions
- Hepatocellular Carcinoma (HCC) at 6-12 Months: Participants with hepatocellular carcinoma (HCC) looking at 18 lesions
Arm/Group | Hepatocellular Carcinoma (HCC) at 6 Weeks | Hepatocellular Carcinoma (HCC) at 6-12 Months
Number analyzed (Participants) | 24 | 7
Number analyzed (lesions) | 25 | 18
lesions
  Stable Disease | 8 | 0
  Partial Response | 6 | 4
  Complete Response | 11 | 14

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- SubStudy 1: Data analysis only for a subset of patients with HCC undergoing hepatic resection compared to healthy controls
- SubStudy 2: Data results only for patients with unresectable HCC treated with Yttrium 90 radioembolization
Arm/Group | Healthy Participant | SubStudy 1 | SubStudy 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 2/32 | 6/24
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/32 | 0/24
Other Adverse Events (participants affected / at risk) | 1/8 | 3/32 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Participant (N=8) | SubStudy 1 (N=32) | SubStudy 2 (N=24)
Mild contrast reaction (General disorders) | 0 | 2 | 0
Unable to tolerate carbogen (Product Issues) | 0 | 1 | 0
Left eye pain (Eye disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT01871545/Prot_SAP_000.pdf